CLINICAL TRIAL: NCT06159205
Title: Investigation of the Effects of Core Stability Exercises Added to the Standard Exercise Program on Patient-Reported and Performance-Based Outcomes in Total Knee Arthroplasty Patients Followed With Telerehabilitation
Brief Title: Core Stability Via Telerehabitation on TKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Burdur Mehmet Akif Ersoy University (Other)
Collaborators: Pamukkale University (Other)
Responsible Party: Principal Investigator, Akın Süzer, Principal Investigator, Burdur Mehmet Akif Ersoy University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ErsoyU.E-60116787-020-90137
Record Dates: First submitted 2023-11-25; First posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Knee Arthropathy; Telerehabilitation
Keywords: total knee arthroplasty; exercise; core stability; telerehabilitation; physiotherapy
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: This study was designed as a double-blind, randomised controlled trial.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: SE Group (Experimental): SE: standard exercises During the follow-up period, only the interventions included in the standard exercise program were applied to the SE Group.
  Interventions: Other: standard exercises
- Group 2: SE + CSE Group (Experimental): CSE: core stability exercises During the follow-up period interventions included in both the standard and core stability program were applied to the SE + CSE group.
  Interventions: Other: standard exercises; Other: core stability exercises

INTERVENTIONS:
Other: standard exercises — Standard exercises for TKA patients.
Other: core stability exercises — Core stability exercises for TKA patients.
  Arms: Group 2: SE + CSE Group

SUMMARY:
Objective: To investigate the effects of core stability exercises (CSE) added to the standard exercises (SE) on patient-reported (PR) and performance-based (PB) outcomes in patients with total knee arthroplasty (TKA) followed with telerehabilitation (TR).

Methods: The 42 patients who participated in the study were randomly divided into 2 groups [group 1: SE (n= 21), group 2: SE + CSE (n= 21)]. The first 8 weeks of the post-discharge follow-up were performed by videoconference-based TR under the supervision of a physiotherapist and the last 4 weeks by telephone-based TR. Functional level was assessed by Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), pain intensity by Visual Analog Scale (VAS), affected knee range of motion (ROM) by Copenhagen Knee Range of Motion Scale (CKRS), quality of life by Short Form-12 (SF-12) and World Health Organization Quality of Life Scale Brief Version (WHOQOL-BREF), lower extremity muscle strength by 30-seconds Chair-Stand Test and locomotor performance by Stair Climb Test. Assessments were performed with TR preoperatively and at the first, second and third post-op months.

DETAILED DESCRIPTION:
At the beginning of the study, an exercise booklet and exercise videos were prepared to be followed throughout the follow-up period. Subsequently, a telerehabilitation (TR) system was established using a laptop computer, a smartphone and a camera as hardware and WhatsApp® and Zoom® applications as software. The surgeries of all patients participating in the study were performed by the same surgical team with fast-track surgical procedure. Until discharge (1 day), a standard physiotherapy and rehabilitation (PTR) program consisting of range of motion and strengthening exercises, cold application, weight transfer and walking training was applied to both groups of patients. At the time of discharge, each patient was given an exercise booklet according to the intervention group.

During the follow-up period, only the interventions included in the standard exercise (SE) program were applied to the SE group, while interventions included in both the SE and core stability exercise (CSE) program were applied to the SE + CSE group. In addition to the TR sessions, each patient performed the interventions belonging to the group they were included in as a home program (HP), 3 sessions per day for the first 8 weeks of the follow-up period. Patient follow-up, which started from the 1st week after discharge, continued for 12 weeks. The content of the follow-up process was planned to include information, assessment, and PTR interventions. The first 8 weeks of the follow-up period consisted of PTR sessions performed with video-conference-based TR method under the supervision of a physiotherapist and HP, while the last 4 weeks consisted of the follow-up of the walking program performed with telephone-based TR method.

ELIGIBILITY:
Inclusion Criteria:

* To be over 18 years old
* Undergoing primary unilateral TKA
* To be able to understand, speak and write Turkish,
* be able to understand verbal and written information, have internet access
* be able to use a video conferencing program

Exclusion Criteria:

* To undergo revision TKA
* To have undergone any major surgery on the lower extremities
* Comorbid diseases such as rheumatoid arthritis, cancer, etc,
* Neurological disease causing functional disability
* Have a diagnosed psychiatric disorder
* Being addicted to alcohol or drugs
* Have a hearing or visual impairment that cannot be corrected with hearing aids or glasses,
* Being morbidly obese (BMI>40 kg/m2)
* be unable to participate in a twelve-week rehabilitation program

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-02-17 (Actual); Study Completion 2023-02-17 (Actual)

PRIMARY OUTCOMES:
Functional level | The assessments were performed before surgery and at the first, second and third months after surgery.
  Functional level was assessed using the Western Ontario McMaster University Osteoarthritis Index. Western Ontario and McMaster Universities Osteoarthritis Index consists of 24 questions and 3 subcategories (pain, stiffness and physical function). Pain is evaluated with 5 questions, stiffness with 2 questions and physical function with 17 questions. Each question in the Index is scored from 0 (none) to 4 (very severe, very difficult). The total score can be a minimum of 0 and a maximum of 100. In addition, each subcategory can also be evaluated on its own. A higher score on the Index indicates more symptoms and physical disability.
Pain intensity | The assessments were performed before surgery and at the first, second and third months after surgery.
  Pain intensity was assessed using the pain subcategory of Western Ontario McMaster University Osteoarthritis Index and the Visual Analog Scale. There are 5 questions in the pain subcategory of the Western Ontario and McMaster Universities Osteoarthritis Index. Each question in the Index is scored from 0 (none) to 4 (very severe, very difficult). The pain score can be a minimum of 0 and a maximum of 20. A higher pain score indicates more pain. Visual Analog Scale consists of a horizontal 10 cm straight line. When viewed from left to right, there is a value of 0 at the beginning and 10 at the end of the line. The 0 point of the line indicates no pain and the 10 point indicates the most severe pain felt in life.
Knee range of motion | The assessments were performed before surgery and at the first, second and third months after surgery.
  Knee range of motion was assessed using the Copenhagen Knee Range of Motion Scale. In this scale, knee range of motion is assessed based on illustrations. For the knee joint flexion angle, 6 different illustrations are used: 60°, 75°, 90°, 105°, 120° and 135°. For the knee extension angle, 5 different illustrations are used: 45°, 30°, 15°, 0° and -15°.
Health-related quality of life | The assessments were performed before surgery and at the first, second and third months after surgery.
  Health-related quality of life was assessed with the Short Form-12. In the Short Form-12, the physical component summary-12 score is obtained from the physical functioning, physical role, body pain and general health sub-dimensions, while the mental component summary-12 score is obtained from the vitality, social functioning, emotional role and mental health sub-dimensions. Both physical component summary-12 and mental component summary-12 scores range between 0-100, with higher scores indicating better health status.
General quality of life | The assessments were performed before surgery and at the first, second and third months after surgery.
  General quality of life was assessed with the World Health Organization Quality of Life Brief Version. World Health Organization Quality of Life Brief Version consists of 4 domains: physical health, psychological, social relationships and environment. In World Health Organization Quality of Life Brief Version, each domain is scored separately and expressed as a percentage between 0 and 100, with a higher percentage indicating better health.
Lower extremity muscle strength | The assessments were performed before surgery and at the first, second and third months after surgery.
  Lower extremity muscle strength was assessed with the 30-seconds chair-stand test. The number of times the patient stands up completely from the chair within 30 seconds is recorded as the patient's score.
Locomotor performance | The assessments were performed before surgery and at the first, second and third months after surgery.
  Locomotor performance was assessed with the stair climb test. The time taken to ascend and then descend a 9-step staircase was recorded as the patient's score.

CONTACTS AND LOCATIONS:
Overall Officials: Akın Süzer, PT, PhD, Principal Investigator — Burdur Mehmet Akif Ersoy University; Nihal Büker, PT, PhD, Study Director — Pamukkale University; Harun R Güngör, MD, PhD, Principal Investigator — Pamukkale University; Nusret Ök, MD, PhD, Principal Investigator — Pamukkale University; Raziye Şavkın, PT, PhD, Principal Investigator — Pamukkale University
Locations (2):
- Turkey (Türkiye) (2):
  - Burdur Mehmet Akif Ersoy University, Burdur
  - Pamukkale University, Denizli

IPD SHARING:
Plan to Share IPD: No